CLINICAL TRIAL: NCT01859312
Title: A Pilot Study Assessing the Use of Continuous Subcutaneous Hydrocortisone Infusion in the Treatment of Congenital Adrenal Hyperplasia
Brief Title: Comparison of Cortisol Pump With Standard Treatment for Congenital Adrenal Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130121; 13-CH-0121 (Other: National Institute of Child Health and Human Development)
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-10-02

CONDITIONS: Adrenal Insufficiency; Excess Androgen; Congenital Adrenal Hyperplasia (CAH)
Keywords: Glucocorticoids; Adrenal Insufficiency; Congenital Adrenal Hyperplasia (CAH); Adrenal
MeSH Terms: conditions — Adrenal Insufficiency; Hyperandrogenism; Adrenal Hyperplasia, Congenital | interventions — Hydrocortisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Continuous Subcutaneous Hydrocortisone Infusion (Experimental): Enrolled participants with congenital adrenal hyperplasia (CAH) received continuous subcutaneous hydrocortisone (Solucortef) infusion (CSHI) via insulin pump (Medtronic) (MMT-722Na) to achieve near-physiologic cortisol replacement therapy. Participants were their own controls; participant's baseline outcomes/lab values while on conventional glucocorticoid therapy were compared to outcomes/lab values after 6 months of treatment using CSHI via insulin pump.
  Interventions: Drug: Hydrocortisone (Solucortef); Device: Insulin pump (Medtronic)

INTERVENTIONS:
Drug: Hydrocortisone (Solucortef) — Continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722NA). Total daily hydrocortisone dose was calculated based on the patient's estimated cortisol clearance. Rates were established to achieve peak and trough concentrations within the normal circadian cortisol range.
  Other Names: CSHI
Device: Insulin pump (Medtronic) — Continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722NA)
  Other Names: CSHI

SUMMARY:
Background:

* Congenital adrenal hyperplasia (CAH) is a genetic disorder of the adrenal gland. The adrenal gland is located in the abdomen and produces small amounts of hormones such as cortisol, aldosterone, and androgen. These hormones help control blood pressure, protect the body, and maintain good health, especially during development. People with CAH do not make enough cortisol and aldosterone, and make too much androgen. This can lead to serious medical problems. The standard treatment is to take pills that mimic the effects of cortisol and aldosterone. However, treatment with pills can have long-term side effects because of the higher doses needed, and may not work well for some people.
* A possible new treatment for CAH is to use a pump to deliver cortisol under the skin. Similar pumps are often used to give insulin to people with diabetes. Researchers think that a cortisol pump might be able to help the body use the cortisol more effectively than taking pills. They want to compare the results of a cortisol pump and standard pill treatments for CAH.

Objectives:

- To compare the effectiveness of a cortisol pump with standard cortisol pill therapy for CAH.

Eligibility:

- Men and women at least 18 years of age who have CAH (see more details in Eligibility section below).

Design:

* This study will involve four inpatient hospital stays at the National Institutes of Health in Bethesda, MD over 6 months (spaced 2 months apart). The first and last stays will last about 5 days. The second and third stays will last about 3 days.
* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* At the first study visit, participants will provide regular blood and urine samples. They will also have imaging studies. These studies will look at the bones, fat, and muscles in the abdomen and pelvis.
* Participants will receive a cortisol pump during the first visit. They will be shown how to use the pump. They will also learn what to do, if they need to take extra "stress dose" cortisol pills.
* At the second and third visits, the cortisol dose given with the pump will be adjusted as needed. Blood and urine samples will also be collected. No imaging studies are scheduled for these visits.
* The last study visit will have the same tests as the first visit. Participants will be offered the chance to continue with the pump treatment for 1 more year, or go back to their standard pill treatment.

Study type: Interventional non-randomized trial

Official title: A Pilot Study Assessing the use of Continuous Subcutaneous Hydrocortisone Infusion In the Treatment of Congenital Adrenal Hyperplasia

Estimated enrollment: 8

Study Start Date: May 2013

Estimated Study Completion Date: December 2016

Sponsoring Institute: National Institute of Child Health and Human Development

<TAB>ELIGIBILITY

Inclusion criteria

1. Men and women 18 years of age or older with classic congenital adrenal hyperplasia (21-Hydroxylase deficiency)
2. High adrenal androgens in the blood, and
3. One or more of the following conditions: obesity, fatty liver, risk for diabetes, low bone mass, inability to tolerate cortisol pills

Exclusion criteria

1. Pregnancy
2. Breast feeding
3. Use of inhaled or oral steroids for diseases other than CAH
4. Use of estrogen-containing birth control pills
5. Use of medicines that cross-react with hydrocortisone
6. Use of stress dose steroids for illness during the last 30 days prior to joining the study

DETAILED DESCRIPTION:
Congenital adrenal hyperplasia (CAH) is a common genetic endocrine disorder, with 21-hydroxylase enzyme deficiency accounting for 95% of the cases. 21-hydroxylase deficiency presents with a spectrum of clinical manifestations ranging from salt-wasting and virilization of female neonates (classic CAH) to symptomatic (precocious puberty, short stature, acne) or asymptomatic hyperandrogenemia (non-classic CAH). Classic CAH is characterized by impaired cortisol and mineralocorticoid biosynthesis, which triggers adrenocorticotropic hormone (ACTH) hyper-secretion and accumulation of adrenal androgens. Glucocorticoid treatment of patients with classic CAH focuses on cortisol replacement and prevention of the ACTH-driven androgen excess. Current conventional glucocorticoid treatment regimens (short or long-acting agents dosed once, twice or thrice daily) have failed to simulate physiological cortisol secretion and suppress adrenal androgen overproduction, without supraphysiologic replacement. Short-term overtreatment with glucocorticoids can lead to iatrogenic Cushing syndrome and long-term use has been associated with the development of obesity, visceral adiposity, insulin resistance and osteoporosis. Isolated case reports have provided evidence that continuous subcutaneous hydrocortisone infusion (CSHI) can mimic physiologic cortisol release and lead to improved CAH control at doses similar to or lower than the traditional treatment. This pilot study aims to test the hypothesis that difficult-to-treat adult patients with classic CAH will have better adrenal androgen control and improved CAH and glucocorticoid-related comorbidities, when they receive near-physiologic cortisol replacement therapy via CSHI compared to conventional glucocorticoid treatment. In addition, this study will provide information on the safety and tolerability of CSHI, and will generate data that will be used in the design of future pediatric studies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with known classic CAH due to 21-hydroxylase deficiency as evidenced by hormonal and genetic testing
* Male or female patients 18 years or older
* Females must have a negative pregnancy test initially and at all visits. Sexually active females must be using a medically acceptable method of contraception.
* Patients with elevated adrenal androgens (defined as 17-OHP >1200 ng/dL and androstenedione >210 ng/dL)
* One or more co-morbidities:<TAB>
* Obesity [body mass index (BMI) greater than 30.0 kg/m(2)]
* Fatty liver disease; assessed by AST/ALT liver enzyme ratio (AST to ALT ratio <1 (11)) liver ultrasound or MRI imaging (Steatosis score as previously described)
* Low insulin sensitivity; assessed by the Homeostasis Model Assessment Insulin Resistance (HOMA-IR) method [HOMA-IR = insulin (micro U/ml) times glucose (mmol/L)/ 22.5]. Elevated HOMA-IR index is defined as >2.6 in adults17.
* Osteopenia [bone mineral density by DEXA (at the spine, hip, or forearm) with T-score of -1 to -2.5) or osteoporosis (bone mineral density by DEXA (at the spine, hip, or forearm) with T-score of <-2.5] defined according to World Health Organization (WHO).
* Glucocorticoid-related gastrointestinal side effects (nausea, vomiting, dyspepsia, anorexia, gastritis, peptic ulcer disease and gastric bleeding)

EXCLUSION CRITERIA:

* Co-morbid conditions requiring daily administration of medications that induce hepatic enzymes or interfere with the metabolism of glucocorticoids
* Females who are pregnant or lactating
* Patients on inhaled or oral steroids given for reasons other than treatment of CAH
* Women who have taken estrogen-containing oral contraceptive pills within 6 weeks of recruitment
* Patients who required stress dose glucocorticoids for an illness within 4 weeks of recruitment
* Patients who changed their glucocorticoid agent within 3 months of recruitment
* Patients who underwent bilateral adrenalectomy
* Co-morbid conditions that could interfere with the ability to comply to the protocol

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05-06; Primary Completion 2016-12-02 (Actual); Study Completion 2016-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah P Merke, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Debono M, Ghobadi C, Rostami-Hodjegan A, Huatan H, Campbell MJ, Newell-Price J, Darzy K, Merke DP, Arlt W, Ross RJ. Modified-release hydrocortisone to provide circadian cortisol profiles. J Clin Endocrinol Metab. 2009 May;94(5):1548-54. doi: 10.1210/jc.2008-2380. Epub 2009 Feb 17. PMID 19223520
- [Background] Finkielstain GP, Kim MS, Sinaii N, Nishitani M, Van Ryzin C, Hill SC, Reynolds JC, Hanna RM, Merke DP. Clinical characteristics of a cohort of 244 patients with congenital adrenal hyperplasia. J Clin Endocrinol Metab. 2012 Dec;97(12):4429-38. doi: 10.1210/jc.2012-2102. Epub 2012 Sep 18. PMID 22990093
- [Background] Arlt W, Willis DS, Wild SH, Krone N, Doherty EJ, Hahner S, Han TS, Carroll PV, Conway GS, Rees DA, Stimson RH, Walker BR, Connell JM, Ross RJ; United Kingdom Congenital Adrenal Hyperplasia Adult Study Executive (CaHASE). Health status of adults with congenital adrenal hyperplasia: a cohort study of 203 patients. J Clin Endocrinol Metab. 2010 Nov;95(11):5110-21. doi: 10.1210/jc.2010-0917. Epub 2010 Aug 18. PMID 20719839
- [Result] Nella AA, Mallappa A, Perritt AF, Gounden V, Kumar P, Sinaii N, Daley LA, Ling A, Liu CY, Soldin SJ, Merke DP. A Phase 2 Study of Continuous Subcutaneous Hydrocortisone Infusion in Adults With Congenital Adrenal Hyperplasia. J Clin Endocrinol Metab. 2016 Dec;101(12):4690-4698. doi: 10.1210/jc.2016-1916. Epub 2016 Sep 28. PMID 27680873
- [Derived] Mallappa A, Nella AA, Sinaii N, Rao H, Gounden V, Perritt AF, Kumar P, Ling A, Liu CY, Soldin SJ, Merke DP. Long-term use of continuous subcutaneous hydrocortisone infusion therapy in patients with congenital adrenal hyperplasia. Clin Endocrinol (Oxf). 2018 Oct;89(4):399-407. doi: 10.1111/cen.13813. Epub 2018 Aug 8. PMID 30003563
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-CH-0121.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight adult patients with classic CAH due to 21-hydroxylase deficiency participated in this study. Four were recruited from a pool of 147 patients enrolled on a natural history study at the NIH natural history study (NCT00250159); 4 were recruited through advertisements.
Groups:
- Continuous Sub-Q Hydrocortisone Infusion: Enrolled participants with congenital adrenal hyperplasia (CAH) received continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722Na) to achieve near-physiologic cortisol replacement therapy
  Hydrocortisone (Solucortef): Continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722NA)
  Insulin pump (Medtronic): Continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722NA)
Period: Overall Study
Arm/Group | Continuous Sub-Q Hydrocortisone Infusion
Started | 8
Completed | 8 (Based on medication & supply accountability, one participant was found to be partially non-compliant)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Continuous Sub-Q Hydrocortisone Infusion: Enrolled participants with congenital adrenal hyperplasia (CAH) will receive continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722Na) to deliver near-physiologic cortisol replacement therapy
  Hydrocortisone (Solucortef): Continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722NA)
  Insulin pump (Medtronic): Continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722NA)
Arm/Group | Continuous Sub-Q Hydrocortisone Infusion
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5
  Canada | 3
Phenotype [Count of Participants; unit: Participants]
  Simple Virilizing (SV) | 2
  Salt-wasting (SW) | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With 17-OHP Levels Equal or Below 1,200 ng/dL at 0700
Description: 17-OHP (17-hydroxyprogesterone) is a laboratory blood test to test for congenital adrenal hyperplasia (CAH) due to 21-hydroxylase deficiency
Time Frame: At baseline
Measure: Count of Participants; unit: Participants
Groups:
- Continuous Subcutaneous Hydrocortisone Infusion: Enrolled participants with congenital adrenal hyperplasia (CAH) will receive continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722Na) to deliver near-physiologic cortisol replacement therapy
  Hydrocortisone (Solucortef): Continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722NA)
  Insulin pump (Medtronic): Continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722NA)
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
Participants | 0

2. Primary Outcome: Number of Patients With 17-OH Progesterone Levels Equal or Below 1,200 ng/dL at 0700
Description: as for outcome 1
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
Participants | 3

3. Secondary Outcome: Participants Mean Level of 17-OHP at 0700
Description: as for outcome 1
Time Frame: At baseline
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
ng/dL | 8313 (2748)

4. Secondary Outcome: Participants Mean Level of 17-OHP at 0700
Description: as for outcome 1
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
ng/dL | 2150 (531)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; Comparisons of CSHI (at 6 months) with conventional glucocorticoid therapy (at baseline) were made. Continuous data between baseline and 6 months were compared by paired t tests; Test type: Other; p = 0.021, t-test, 2 sided

5. Secondary Outcome: Participants Mean Level of 17-OHP Area Under the Curve (AUC) - 24 Hours
Description: 17-OHP (17-hydroxyprogesterone) is a laboratory blood test to test for congenital adrenal hyperplasia (CAH) due to 21-hydroxylase deficiency. AUC was calculated using the linear-up log-down trapezoidal rule for the entire 24 hours and samples were obtained every 2 hours beginning at 2300, 0100, 0300, 0500, 0700, 0900, 1100, 1300, 1500, 1700, 1900, 2100, 2300. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 98.5 (39.3)

6. Secondary Outcome: Participants Mean Level of 17-OHP Area Under the Curve (AUC) - 24 Hours
Description: as for outcome 5
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 25.7 (9.5)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.027, t-test, 2 sided

7. Secondary Outcome: Participants Mean Level of 17-OHP Area Under the Curve (AUC) - Daytime (0700-1500)
Description: 17-OHP (17-hydroxyprogesterone) is a laboratory blood test to test for congenital adrenal hyperplasia (CAH) due to 21-hydroxylase deficiency. AUC was calculated using the linear-up log-down trapezoidal rule for the 8 hour daytime level, samples were obtained every 2 hours beginning at 0700, 0900, 1100, 1300, 1500. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 48.6 (22.4)

8. Secondary Outcome: Participants Mean Level of 17-OHP Area Under the Curve (AUC) - Daytime (0700-1500)
Description: as for outcome 7
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 6.8 (1.8)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.008, t-test, 2 sided

9. Secondary Outcome: Participants Mean Level of 17-OHP Area Under the Curve (AUC) - Midday (1500 - 2300)
Description: 17-OHP (17-hydroxyprogesterone) is a laboratory blood test to test for congenital adrenal hyperplasia (CAH) due to 21-hydroxylase deficienc. AUC was calculated using the linear-up log-down trapezoidal rule for the 8 hour midday level, samples were obtained every 2 hours beginning at 1500, 1700, 1900, 2100, 2300. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 20.5 (6.8)

10. Secondary Outcome: Participants Mean Level of 17-OHP Area Under the Curve (AUC) - Midday (1500 - 2300)
Description: 17-OHP (17-hydroxyprogesterone) is a laboratory blood test to test for congenital adrenal hyperplasia (CAH) due to 21-hydroxylase deficiency. AUC was calculated using the linear-up log-down trapezoidal rule for the 8 hour midday level, samples were obtained every 2 hours beginning at 1500, 1700, 1900, 2100, 2300. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 7.5 (4.9)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.012, t-test, 2 sided

11. Secondary Outcome: Participants Mean Level of 17-OHP Area Under the Curve (AUC) - Nighttime (2300 - 0700)
Description: 17-OHP (17-hydroxyprogesterone) is a laboratory blood test to test for congenital adrenal hyperplasia (CAH) due to 21-hydroxylase deficiency. AUC was calculated using the linear-up log-down trapezoidal rule for the 8 hour nighttime level, samples were obtained every 2 hours beginning at 2300, 0100, 0300, 0500, 0700. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 29.5 (11.1)

12. Secondary Outcome: Participants Mean Level of 17-OHP Area Under the Curve (AUC) - Nighttime (2300 - 0700)
Description: as for outcome 11
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 11.4 (3.0)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.157, t-test, 2 sided

13. Secondary Outcome: Participants Mean Level of Androstenedione at 0700
Description: Participants Mean Level of Androstenedione at 0700.
Time Frame: At baseline
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
ng/dL | 748 (295)

14. Secondary Outcome: Participants Mean Level of Androstenedione at 0700
Description: Participants Mean Level of Androstenedione at 0700.
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
ng/dL | 317 (77)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.015, t-test, 2 sided

15. Secondary Outcome: Participants Mean Level of Androstenedione Area Under the Curve (AUC) - 24 Hours
Description: Participants Mean Level of Androstenedione Area Under the Curve (AUC) - 24 hours. AUC was calculated using the linear-up log-down trapezoidal rule for the entire 24 hours and samples were obtained every 2 hours beginning at 2300, 0100, 0300, 0500, 0700, 0900, 1100, 1300, 1500, 1700, 1900, 2100, 2300. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 12.7 (4.5)

16. Secondary Outcome: Participants Mean Level of Androstenedione Area Under the Curve (AUC) - 24 Hours
Description: as for outcome 15
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 5.2 (1.4)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.009, t-test, 2 sided

17. Secondary Outcome: Participants Mean Level of Androstenedione Area Under the Curve (AUC) - Daytime (0700-1500)
Description: Participants Mean Level of Androstenedione Area Under the Curve (AUC) - Daytime (0700-1500). AUC was calculated using the linear-up log-down trapezoidal rule for the 8 hour daytime level, samples were obtained every 2 hours beginning at 0700, 0900, 1100, 1300, 1500. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 5.3 (2.1)

18. Secondary Outcome: Participants Mean Level of Androstenedione Area Under the Curve (AUC) - Daytime (0700-1500)
Description: as for outcome 17
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 1.8 (0.4)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.008, t-test, 2 sided

19. Secondary Outcome: Participants Mean Level of Androstenedione Area Under the Curve (AUC) - Midday (1500 - 2300)
Description: Participants Mean Level of Androstenedione Area Under the Curve (AUC) - Midday (1500 - 2300). AUC was calculated using the linear-up log-down trapezoidal rule for the 8 hour midday level, samples were obtained every 2 hours beginning at 1500, 1700, 1900, 2100, 2300. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 3.7 (1.1)

20. Secondary Outcome: Participants Mean Level of Androstenedione Area Under the Curve (AUC) - Midday (1500 - 2300)
Description: as for outcome 19
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 1.6 (0.6)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.009, t-test, 2 sided

21. Secondary Outcome: Participants Mean Level of Androstenedione Area Under the Curve (AUC) - Nighttime (2300 - 0700)
Description: Participants Mean Level of Androstenedione Area Under the Curve (AUC) - Nighttime (2300 - 0700). AUC was calculated using the linear-up log-down trapezoidal rule for the 8 hour nighttime level, samples were obtained every 2 hours beginning at 2300, 0100, 0300, 0500, 0700. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 3.7 (1.3)

22. Secondary Outcome: Participants Mean Level of Androstenedione Area Under the Curve (AUC) - Nighttime (2300 - 0700)
Description: as for outcome 21
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*mcg/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*mcg/dL | 1.8 (0.4)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.043, t-test, 2 sided

23. Secondary Outcome: Participants Mean Level of ACTH at 0700
Description: Participants Mean Level of ACTH at 0700.
Time Frame: At baseline
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
pg/mL | 405 (114)

24. Secondary Outcome: Participants Mean Level of ACTH at 0700
Description: Participants Mean Level of ACTH at 0700.
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
pg/mL | 139 (47)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.024, t-test, 2 sided

25. Secondary Outcome: Participants Mean Level of ACTH Area Under the Curve (AUC) - 24 Hours
Description: Participants Mean Level of ACTH Area Under the Curve (AUC) - 24 Hours. AUC was calculated using the linear-up log-down trapezoidal rule for the entire 24 hours and samples were obtained every 2 hours beginning at 2300, 0100, 0300, 0500, 0700, 0900, 1100, 1300, 1500, 1700, 1900, 2100, 2300.Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*pg/mL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*pg/mL | 2538 (743)

26. Secondary Outcome: Participants Mean Level of ACTH Area Under the Curve (AUC) - 24 Hours
Description: Participants Mean Level of ACTH Area Under the Curve (AUC) - 24 Hours. AUC was calculated using the linear-up log-down trapezoidal rule for the entire 24 hours and samples were obtained every 2 hours beginning at 2300, 0100, 0300, 0500, 0700, 0900, 1100, 1300, 1500, 1700, 1900, 2100, 2300. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*pg/mL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*pg/mL | 1087 (359)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.031, t-test, 2 sided

27. Secondary Outcome: Participants Mean Level of ACTH Area Under the Curve (AUC) - Daytime (0700-1500)
Description: Participants Mean Level of ACTH Area Under the Curve (AUC) - Daytime (0700-1500). AUC was calculated using the linear-up log-down trapezoidal rule for the 8 hour daytime level, samples were obtained every 2 hours beginning at 0700, 0900, 1100, 1300, 1500. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*pg/mL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*pg/mL | 1239 (402)

28. Secondary Outcome: Participants Mean Level of ACTH Area Under the Curve (AUC) - Daytime (0700-1500)
Description: as for outcome 27
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*pg/mL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*pg/mL | 340 (107)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.005, t-test, 2 sided

29. Secondary Outcome: Participants Mean Level of ACTH Area Under the Curve (AUC) - Midday (1500 - 2300)
Description: Participants Mean Level of ACTH Area Under the Curve (AUC) - Midday (1500 - 2300). AUC was calculated using the linear-up log-down trapezoidal rule for the 8 hour midday level, samples were obtained every 2 hours beginning at 1500, 1700, 1900, 2100, 2300. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*pg/mL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*pg/mL | 458 (179)

30. Secondary Outcome: Participants Mean Level of ACTH Area Under the Curve (AUC) - Midday (1500 - 2300)
Description: as for outcome 29
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*pg/mL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*pg/mL | 183 (55)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.004, t-test, 2 sided

31. Secondary Outcome: Participants Mean Level of ACTH Area Under the Curve (AUC) - Nighttime (2300 - 0700)
Description: Participants Mean Level of ACTH Area Under the Curve (AUC) - Nighttime (2300 - 0700). AUC was calculated using the linear-up log-down trapezoidal rule for the 8 hour nighttime level, samples were obtained every 2 hours beginning at 2300, 0100, 0300, 0500, 0700. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*pg/mL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*pg/mL | 841 (233)

32. Secondary Outcome: Participants Mean Level of ACTH Area Under the Curve (AUC) - Nighttime (2300 - 0700)
Description: as for outcome 31
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*pg/mL
Groups:
- Continuous Subcutaenous Hydrocortisone Infusion: Enrolled participants with congenital adrenal hyperplasia (CAH) will receive continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722Na) to deliver near-physiologic cortisol replacement therapy
  Hydrocortisone (Solucortef): Continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722NA)
  Insulin pump (Medtronic): Continuous subcutaneous hydrocortisone infusion (CSHI) via Medtronic insulin pump (MMT-722NA)
Arm/Group | Continuous Subcutaenous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*pg/mL | 564 (216)
Statistical Analysis 1: Comparison: Continuous Subcutaenous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.524, t-test, 2 sided

33. Secondary Outcome: Participants Mean Progesterone Levels at 0700
Description: Participants Mean Level of Progesterone at 0700
Time Frame: At baseline
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
ng/mL | 9.5 (5.4)

34. Secondary Outcome: Participants Mean Progesterone Level at 0700
Description: Participants Mean Level of Progesterone at 0700
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
ng/mL | 0.8 (0.4)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.007, t-test, 2 sided; Comparison of hormone levels on conventional glucocorticoid therapy at baseline and following 6 months of CSHI

35. Secondary Outcome: Participants Mean Level of Progesterone Area Under the Curve (AUC) - 24 Hours
Description: Participants Mean Level of Progesterone area under the curve (AUC) - 24 hours. AUC was calculated using the linear-up log-down trapezoidal rule for the entire 24 hours and samples were obtained every 2 hours beginning at 2300, 0100, 0300, 0500, 0700, 0900, 1100, 1300, 1500, 1700, 1900, 2100, 2300. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*ng/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*ng/dL | 101.1 (48.8)

36. Secondary Outcome: Participants Mean Level of Progesterone Area Under the Curve (AUC) - 24 Hours
Description: as for outcome 35
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*ng/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*ng/dL | 13.7 (4.6)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.084, t-test, 2 sided

37. Secondary Outcome: Participants Mean Level of Progesterone Area Under the Curve (AUC) - Daytime (0700-1500)
Description: Participants Mean Level of Progesterone area under the curve (AUC) - Daytime (0700-1500). AUC was calculated using the linear-up log-down trapezoidal rule for the 8 hour daytime level, samples were obtained every 2 hours beginning at 0700, 0900, 1100, 1300, 1500. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*ng/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*ng/dL | 42.2 (20.0)

38. Secondary Outcome: Participants Mean Level of Progesterone Area Under the Curve (AUC) - Daytime (0700-1500)
Description: as for outcome 37
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*ng/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*ng/dL | 4.2 (1.6)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.057, t-test, 2 sided

39. Secondary Outcome: Participants Mean Level of Progesterone Area Under the Curve (AUC) - Midday (1500 - 2300)
Description: Participants Mean Level of Progesterone area under the curve (AUC) - Midday (1500 - 2300). AUC was calculated using the linear-up log-down trapezoidal rule for the 8 hour midday level, samples were obtained every 2 hours beginning at 1500, 1700, 1900, 2100, 2300. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*ng/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*ng/dL | 30.7 (17.7)

40. Secondary Outcome: Participants Mean Level of Progesterone Area Under the Curve (AUC) - Midday (1500 - 2300)
Description: as for outcome 39
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*ng/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*ng/dL | 5.5 (3.2)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.103, t-test, 2 sided

41. Secondary Outcome: Participants Mean Level of Progesterone Area Under the Curve (AUC) - Nighttime (2300 - 0700)
Description: Participants Mean Level of Progesterone area under the curve (AUC) - Nighttime (2300 - 0700). AUC was calculated using the linear-up log-down trapezoidal rule for the 8 hour nighttime level, samples were obtained every 2 hours beginning at 2300, 0100, 0300, 0500, 0700. Actual collection times were used to define peak plasma concentration (Cmax) and time to peak plasma concentration (Tmax).
Time Frame: At baseline
Measure: Mean (Standard Error); unit: h*ng/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*ng/dL | 28.2 (12.5)

42. Secondary Outcome: Participants Mean Level of Progesterone Area Under the Curve (AUC) - Nighttime (2300 - 0700)
Description: as for outcome 41
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: h*ng/dL
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
h*ng/dL | 4.0 (0.5)
Statistical Analysis 1: Comparison: Continuous Subcutaneous Hydrocortisone Infusion; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.070, t-test, 2 sided

43. Secondary Outcome: Participant Lean Body Mass
Description: lean body mass measured by DEXA, Hologic Discovery-A
Time Frame: At baseline
Measure: Mean (Standard Error); unit: kg
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
kg | 60.7 (3.7)

44. Secondary Outcome: Participant Lean Body Mass
Description: lean body mass measured by DEXA, Hologic Discovery-A
Time Frame: At 6 months
Measure: Mean (Standard Error); unit: kg
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
Number analyzed (Participants) | 8
kg | 64.3 (4.4)

ADVERSE EVENTS:
Time Frame: At 6 months. Subjects that select the option of continuing CSHI therapy for 1 additional year will be monitored for 1 year, 6 months.
Description: IRB granted a waiver of reporting the following anticipated adverse events (non-UP adverse events) unless they occurring in greater frequency than expected:
  1. Local skin reaction (50%)
  2. Local skin infection requiring local or antibiotic treatment (10%)
  3. Minimal bleeding after removal of the infusion set (90%)
Arm/Group | Continuous Subcutaneous Hydrocortisone Infusion
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Subcutaneous Hydrocortisone Infusion (N=8)
Skin erythema with pruritis at the infusion set site (Skin and subcutaneous tissue disorders) | 3
Local skin infection at the infusion set site (Skin and subcutaneous tissue disorders) | 5
Dizziness (Nervous system disorders) | 5
Lightheadedness (Nervous system disorders) | 5
Weakness (Musculoskeletal and connective tissue disorders) | 3
Fatigue (General disorders) | 7
Nausea (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 7
Carpal tunnel (Musculoskeletal and connective tissue disorders) | 1
Knee pain when walking (Musculoskeletal and connective tissue disorders) | 1
Tinnutus (Ear and labyrinth disorders) | 1
Decreased appetite (Gastrointestinal disorders) | 2
Increased appetite (Gastrointestinal disorders) | 6
Difficulty falling asleep or frequent wakening (General disorders) | 5
Early morning wakening (General disorders) | 3
Increased acne (Skin and subcutaneous tissue disorders) | 2
Weight gain (General disorders) | 5

LIMITATIONS AND CAVEATS:
All patients completed the study; according to medication and supply accountability, one patient was found to be partially non-compliant, the pump was disconnected approximately 30% of the time. When this patient was excluded, analysis were the same.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes